CLINICAL TRIAL: NCT01255904
Title: A RANDOMIZED CONTROLLED TRIAL OF ORAL CHLORAL HYDRATE VERSUS INTRANASAL DEXMEDETOMIDINE FOR SEDATED ABR EXAMS.
Brief Title: A Trial Of Oral Chloral Hydrate Versus Intranasal Dexmedetomidine For Sedated Abr Exams
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Jason Reynolds, Assistant Professor of Pediatrics, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-27453
Record Dates: First submitted 2010-11-18; First posted 2010-12-08 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Sedation
MeSH Terms: interventions — Chloral Hydrate; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Oral Chloral and intranasal placebo
  Interventions: Drug: Chloral Hydrate; Other: Intranasal placebo
- Arm 2 (Experimental): oral placebo and intranasal dexmedetomidine
  Interventions: Drug: Dexmedetomidine; Other: Oral placebo

INTERVENTIONS:
Drug: Chloral Hydrate — Oral chloral hydrate 50 mg/kg
  Arms: Arm 1
Drug: Dexmedetomidine — Intranasal dexmedetomidine 3 mcg/kg
  Arms: Arm 2
Other: Oral placebo — Oral saline administered
  Arms: Arm 2
Other: Intranasal placebo — Intranasal saline administered
  Arms: Arm 1

SUMMARY:
The purpose of this study is to compare the efficacy of oral chloral hydrate to intranasal dexmedetomidine for the successful completion of a sedated ABR exam (hearing exam).

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for ABR exam with sedation to be administered according to protocol by nurse in keeping with standard practice at the TCH Audiology clinic.

Exclusion Criteria:

* Patients younger than 6 months or older than 8 years
* Previously failed sedation
* Weight greater than 25 kg
* Weight less than 5 kg
* BMI above 30
* Diagnosis of ADHD
* Any patient deemed inappropriate for nurse administered sedation
* Patients with any cardiac disease
* Obstructive sleep apnea

Ages: 6 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2011-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Childrens Hospital, Houston, Texas, United States

REFERENCES:
- [Derived] Fong CY, Lim WK, Li L, Lai NM. Chloral hydrate as a sedating agent for neurodiagnostic procedures in children. Cochrane Database Syst Rev. 2021 Aug 16;8(8):CD011786. doi: 10.1002/14651858.CD011786.pub3. PMID 34397100

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Placebo and Intransal Dexmedetomidine: Oral placebo followed by Intranasal dexmedetomidine 3 mcg/kg (max dose 100 mcg).
- Oral Chloral Hydrate and Intranasal Placebo: 50 mg/kg oral chloral hydrate followed by intranasal placebo.
Period: Overall Study
Arm/Group | Oral Placebo and Intransal Dexmedetomidine | Oral Chloral Hydrate and Intranasal Placebo
Started | 45 | 45
Completed | 44 | 41
Not Completed | 1 | 4
Not completed — Physician Decision | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Placebo and Intransal Dexmedetomidine | Oral Chloral Hydrate and Intranasal Placebo | Total
Number analyzed (Participants) | 44 | 41 | 85
Age, Continuous [Mean (Standard Deviation); unit: months] | 23.33 (12.63) | 25.55 (11.21) | 24.40 (11.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 14 | 35
  Male | 23 | 27 | 50
Region of Enrollment [Number; unit: participants]
  United States | 44 | 41 | 85

OUTCOME MEASURES:

1. Primary Outcome: Time to Complete Study
Description: Time from medication administration to study completion.
Time Frame: 60-180 minutes
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Oral Placebo and Intransal Dexmedetomidine | Oral Chloral Hydrate and Intranasal Placebo
Number analyzed (Participants) | 44 | 41
Minutes | 85.5 [80 to 110] | 110 [85 to 119]

ADVERSE EVENTS:
Arm/Group | Oral Placebo and Intransal Dexmedetomidine | Oral Chloral Hydrate and Intranasal Placebo
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/41
Other Adverse Events (participants affected / at risk) | 2/44 | 0/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Placebo and Intransal Dexmedetomidine (N=44) | Oral Chloral Hydrate and Intranasal Placebo (N=41)
mild hypoxia < 94% and > 90% (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
partial airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was not designed to detect small differences in rare adverse and the overall safety of either medication cannot be assessed based on these results alone.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes